CLINICAL TRIAL: NCT06677541
Title: Vibrator Use to Improve Sexual and Pelvic Floor Function Among Urogynecology Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol 7076
Record Dates: First submitted 2024-10-21; First posted 2024-11-06 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Floor Dysfunction; Sexual Dysfunction Female; Vibrator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control arm (Active Comparator)
  Interventions: Other: Instructional handout
- Intervention arm (Experimental)
  Interventions: Other: Instructional handout; Device: Vibrator

INTERVENTIONS:
Other: Instructional handout — A handout on how to improve sexual dysfunction/function will be provided
Device: Vibrator — An FDA approved vibrator device to improve sexual function will be provided
  Arms: Intervention arm

SUMMARY:
Limited data exist describing the use and role of vibrators in a urogynecology population and no randomized controlled trials investigating the use of vibrators as a therapeutic tool to enhance sexual and pelvic floor function in urogynecology patients has been conducted. This study aims to evaluate the efficacy of vibrator use in improving sexual and pelvic floor function in urogynecology patients who report sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* • Women aged 18 and over presenting to the urogynecology clinic.

  * Women diagnosed with one of the following urogynecologic conditions

    o Pelvic organ prolapse, urgency incontinence, overactive bladder, stress urinary incontinence, fecal incontinence, recovering from a urogynecologic surgery over 6 weeks following surgery and clear for intercourse. Patients post op who continue to have pelvic floor dysfunction can be candidates for the study if they continue to have one of the pelvic floor dysfunctions listed.
  * Patient will be screened with the FSFI and will be eligible if they score less than 26.55
  * Patient's must be willing to use a vibrator.
  * Able to provide informed consent.
  * Not currently using a vibrator or has not used a vibrator in the past 3 months.
  * Able to read and write in English

Exclusion Criteria:

* • Patients with cognitive impairment.

  * Patients with refusal or discomfort with vibrator use.
  * Currently using a vibrator or has used a vibrator in the past 3 months.
  * Patients unable to provide informed consent.
  * Patients not clear for intercourse following their surgery
  * Patients with surgery within 2 months of recruitment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index | up to 12 weeks
  A 19 question validated survey on sexual function with lower scores indicating worse outcome

SECONDARY OUTCOMES:
Pelvic Floor Distress Inventory -20 | up to 12 weeks
  20 question validated survey on pelvic floor dysfunction with lower scores indicating worse outcomes
Pelvic Organ Prolapse incontinence sexual questionnaire 12 | up to 12 weeks
  a 12 question validated survey on sexual function in patients with pelvic floor dysfunction with lower scores indicating worse outcomes
sexual satisfaction index | up to 12 weeks
  a validated questionnaire on sexual satisfaction with lower scores indicating worse outcomes
female genitourinary pain index | up to 12 weeks
  validated survey on genitourinary pain in females with lower scores indicating worse outcomes
patient health questionnaire 9 | up to 12 weeks
  validated questionnaire on depression with lower scores indicating worse outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Uncertain, might be with publication